CLINICAL TRIAL: NCT03787147
Title: Assessing the Efficacy of Virtual Reality Analgesia (VRA) in Adult Patients for Pain Control During Spinal Injections (SI)
Acronym: VR adult
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Never started the study cause of the lack of funding
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Sayed Wahezi, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-9613
Record Dates: First submitted 2018-12-05; First posted 2018-12-26 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: Virtual Reality; Spinal Injection; Adult; Analgesia; Google cardboard; Oculus
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The sealed envelope is randomized and blinded so no one will know which group the participant falls and its revealed only after the participant opens the sealed envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Spinal Injection (Other): Adults receiving Spinal Injection(SI) without Virtual Reality(VR).
  Interventions: Drug: Lidocaine Hydrochloride; Drug: Bupivacaine
- Google Cardboard (Active Comparator): Adults receiving SI while using Google Cardboard Virtual reality head mounted display powered by a iPod touch
  Interventions: Device: Google Cardboard; Drug: Lidocaine Hydrochloride; Drug: Bupivacaine
- Oculus (Active Comparator): Adults receiving SI while using VR with Oculus Rift.
  Interventions: Device: Oculus; Drug: Lidocaine Hydrochloride; Drug: Bupivacaine

INTERVENTIONS:
Device: Google Cardboard — Assessing the Efficacy of Virtual Reality Analgesia (VRA) in Adult Patients for Pain Control During Spinal Injections (SI). VRA is a the oculus or the google cardboard that helps decrease anxiety. The participant in the oculus or the Google cardboard arms are asked to watch VR videos during the spinal injection.
  Arms: Google Cardboard
Device: Oculus — Assessing the Efficacy of Virtual Reality Analgesia (VRA) in Adult Patients for Pain Control During Spinal Injections (SI). VRA is a the oculus or the google cardboard that helps decrease anxiety. The participant in the oculus or the Google cardboard arms are asked to watch VR videos during the spinal injection.
  Arms: Oculus
Drug: Lidocaine Hydrochloride — All groups will receive pharmaceutical analgesia, either lidocaine or bupivacaine, depending on the condition. Dosage and frequency of pharmaceutical analgesia will be tailored to each participant's condition.
Drug: Bupivacaine — All groups will receive pharmaceutical analgesia, either lidocaine or bupivacaine, depending on the condition. Dosage and frequency of pharmaceutical analgesia will be tailored to each participant's condition.

SUMMARY:
A three-group parallel randomized controlled trial to evaluate the efficacy of virtual reality analgesia (VRA) to decrease patient procedural pain and anxiety in the Adult patients undergoing Spinal Injections (SI).

ELIGIBILITY:
Inclusion Criteria:

* Adult requiring Spinal Injections
* Adult > 18years
* Adults with intact vision who can attend VR intervention

Exclusion Criteria:

* Anyone < 18 years
* Adults who are not attentive to VR secondary to poor concentration, poor cognition to external stimuli
* Adults who request moderate IV sedation
* Adults with photic-induced seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity as measured by the Visual Analog Scale | Immediately after receiving spinal injection
  Participants are asked to rate their intensity of pain, by completing a Visual Analog Scale (VAS). The VAS consists of lines and emojis used to indicate pain level; the lines range from 0 (= no pain) to 10 (= unbearable pain) and the emojis range from 0 (= no pain) to 5 (= unbearable pain).

SECONDARY OUTCOMES:
Anxiety Level as measured by the Visual Facial Anxiety Scale | Immediately after receiving spinal injection
  Participants are asked to rate their anxiety level by completing the Visual Facial Anxiety Scale(VFAS). The VFAS consists of emojis ranging from 0 (= no anxiety) to 5 (highest anxiety).
Heart rate as measured by the Empatica E4 wristband | Baseline, during and Immediately after the procedure
  The Empatica E4 wristband is a wearable research device that offers real-time physiological data acquisition and software for in-depth analysis and visualization. Empatica E4 wristband is worn by the participant throughout the procedure to measure heart rate before, during and after the procedure.
Systolic Blood Pressure as measured by the Empatica E4 wristband | Baseline, during and Immediately after the procedure
  The Empatica E4 wristband is a wearable research device that offers real-time physiological data acquisition and software for in-depth analysis and visualization. Empatica E4 wristband is worn by the participant throughout the procedure to measure Blood Pressure before, during and after the procedure.
Diastolic Blood Pressure as measured by the Empatica E4 wristband | Baseline, during and Immediately after the procedure
  The Empatica E4 wristband is a wearable research device that offers real-time physiological data acquisition and software for in-depth analysis and visualization. Empatica E4 wristband is worn by the participant throughout the procedure to measure Blood Pressure before, during and after the procedure.
Sympathetic skin response as measured by the Empatica E4 wristband | Baseline, during and Immediately after the procedure
  The Empatica E4 wristband is a wearable research device that offers real-time physiological data acquisition and software for in-depth analysis and visualization. Empatica E4 wristband is worn by the participant throughout the procedure to measure Sympathetic skin response before, during and after the procedure.
Temperature as measured by the Empatica E4 wristband | Baseline, during and Immediately after the procedure
  The Empatica E4 wristband is a wearable research device that offers real-time physiological data acquisition and software for in-depth analysis and visualization. Empatica E4 wristband is worn by the participant throughout the procedure to measure Temperature before, during and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Wahezi, MD, Principal Investigator — Albert Einstein College of Medicine

IPD SHARING:
Plan to Share IPD: No